CLINICAL TRIAL: NCT05577754
Title: A Phase II Double-blind Multi-center, Placebo-controlled Trial, to Assess the Efficacy and Safety of Alpelisib (BYL719) in Pediatric and Adult Patients With Megalencephaly-CApillary Malformation Polymicrogyria Syndrome (MCAP)
Brief Title: Assessment of the Efficacy and Safety of Alpelisib (BYL719) in Pediatric and Adult Patients With Megalencephaly-CApillary Malformation Polymicrogyria Syndrome (MCAP)
Acronym: SESAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLIVIER FAIVRE Novartis 2021
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Megalencephaly-capillary Malformation Polymicrogyria Syndrome (MCAP)
Keywords: Neurodevelopmental disorders; alpelisib; therapeutic trial; PIK3CA; MCAP
MeSH Terms: conditions — Megalencephaly cutis marmorata telangiectatica congenita; Neurodevelopmental Disorders; Hereditary Sensory and Autonomic Neuropathies | interventions — Alpelisib; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator)
  Interventions: Drug: Alpelisib (BYL719); Drug: Matching placebo; Procedure: Optional lumbar puncture + blood sample
- Group B (Experimental)
  Interventions: Drug: Alpelisib (BYL719); Procedure: Optional lumbar puncture + blood sample

INTERVENTIONS:
Drug: Alpelisib (BYL719) — Administration during open label and double-blind period of group B: alpelisib will be taken once a day each day over 24 mois During open label period of group A: alpelisib will be taken once a day each day over 24 months
Drug: Matching placebo — During double-blind period of group A: matching placebo will be taken once a day each day over 6 months
  Arms: Group A
Procedure: Optional lumbar puncture + blood sample — Between 6 and 24 months of treatment with Alpelisib

SUMMARY:
This study is a two periods multi-center Phase II trial, with a 6 months double-blind, placebo-controlled period followed by open label period, to assess the efficacy and safety of alpelisib (BYL719) in pediatric and adult patients with Megalencephaly-CApillary malformation Polymicrogyria syndrome (MCAP)

DETAILED DESCRIPTION:
This study consists of a screening period up to 90 days, a first double-blind, placebo-controlled period of 6 months, followed by an open label period of alpelisib treatment, to reach a 24-month duration of treatment for all patients. The study will enroll 18-40 years old adults and 2-18 years old paediatric patients.

Eligible patients will be randomized in a 1:1 ratio for the first period (alpelisib or placebo). A first assessment will be performed at 6 months. Patients completing this first period will enter the open label period, and either start alpelisib if they were on placebo, continue at the same dose if responders, or increase dose if not responders (dose increase only possible for children of 5 years old and over), and if no unacceptable toxicity occurs.

Patients will be followed monthly in local centres, and centrally assessed (clinical, biological, neuropsychological and functional evaluation) at baseline and every 6 months. Patients will be evaluated by volumetric MRI at baseline and at 24 months.

Participant may be discontinued from treatment with alpelisib earlier due to unacceptable toxicity, confirmed disease progression, death, and/or any other reason at the discretion of the investigator or the participant.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and assent (when applicable) from the patient, parent, or guardian must be obtained prior to any study related screening procedures are performed.
2. Male or female patients age ≥2 years and ≤40 years at the time of informed consent
3. Patients with diagnosis of MCAP* with neurodevelopmental disorder presentation (from specific learning disorder to severe intellectual disability)
4. Documented evidence of a postzygotic or constitutional mutation(s) in the PIK3CA gene performed in local laboratories using a Deoxyribonucleic acid (DNA) based validated test at the time of informed consent.
5. Adequate bone marrow and organ function (assessed during the screening visit):

   1. Absolute neutrophil count ≥ 1.5 × 109/L
   2. Platelets ≥ 100 × 109/L
   3. Hemoglobin ≥ 9.0 g/dL (transfusions are allowed)
   4. Calcium (corrected for serum albumin) and magnesium within normal limits or ≤Grade 1 according to NCI-CTCAE version 5.0 if judged clinically not significant by the investigator
   5. Potassium within normal limits.
   6. INR ≤1.5
   7. Creatinine Clearance ≥ 30 mL/min using Modification of Diet in Renal Disease
   8. (MDRD) (≥18 years old) or creatinine-based Bedside Schwartz (˂18 years old) Glomerular filtration rate (GFR) equation
   9. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN.
   10. Total bilirubin< ULN except for patients with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN
   11. Fasting plasma glucose (FPG) ≤ 140 mg/dL (7.7 mmol/L) and Glycosylated hemoglobin (HbA1c) ≤ 6.5% (both criteria have to be met)
   12. Fasting Serum lipase ≤ ULN
6. Able to swallow study drug according to age: tablets, or as drinkable suspension, or granules (under development)
7. For women of child-bearing potential only: negative pregnancy test at screening visit
8. Male patients with sexual partners who are pregnant, possibly pregnant or who could become pregnant should use condoms during sexual intercourse for the duration of the study and for one week following discontinuation of alpelisib.

7. For exploratory study only : signed informed optional consent for lumbar puncture

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for inclusion in this study:

1. Patient previously treated with alpelisib
2. Known impairment of GI function due to concomitant disease that may significantly alter the absorption of the study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection) at time of informed consent.
3. Participant with uncontrolled diabetes mellitus (Type I or II) at time of informed consent.
4. History of hypersensitivity to any drugs or metabolites of PI3K inhibitor or any of the excipients of alpelisib at time of informed consent.
5. Participant with other concurrent severe and/or uncontrolled medical conditions that would, in the treating Physician's judgment, contraindicate administration of alpelisib (e.g., active and/or uncontrolled severe infection, chronic active hepatitis, hepatic impairment Child Pugh score C, immuno-compromised, etc.) at time of informed consent.
6. Female participants of childbearing potential and male participants who do not agree at time of informed consent to abstinence or, if sexually active, unwilling to use a condom and/or a highly effective method of contraception for the duration of the study and for one week following discontinuation of alpelisib. Highly effective contraception methods is one of the following:

   1. Total abstinence: when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
   2. Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks before taking alpelisib. In case of oophorectomy alone, only when the reproductive status of the female has been confirmed by follow-up hormone level assessment
   3. Male sterilization at least 6 months prior to screening. The vasectomized male partner should be the sole partner for that study participant
   4. Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the ICF.
7. Treatment by any mTOR or PI3K-AKT signaling pathway inhibitor within 1 month before inclusion
8. History of prior and or ongoing malignancy (within 5 years before informed consent except radically treated Carcinoma in situ of radically treated basal-cell carcinoma of skin or thyroid gland well differentiated microcarcinoma or Stage 1 Wilms' tumor of a histology other than anaplastic), or ongoing investigations or treatment for malignancy at time of informed consent.
9. Treatment with strong inducers of CYP3A4 and inhibitors of Breast Cancer Resistance Protein (BCRP) that cannot be stopped at least the week prior to the screening
10. Debulking or other major surgery performed within 3 months at time of informed consent
11. Known history of Steven Johnson's syndrome, erythema multiform or toxic epidermal necrolysis at time of informed consent.
12. For participants ≥ 6 years of age: Participants with documented pneumonitis or interstitial lung disease at the time of informed consent and with impaired lung function (e.g., FEV1 (Forced expiratory volume) or DLCO (Diffusing Capacity of the Lung for Carbon Monoxide) ≤ 70% of predicted) that is not related to PROS.
13. For participants between 2 to 5 years of age: Participants with documented or suspicious pneumonitis or interstitial lung disease based on MRI images at time of informed consent.
14. History of acute pancreatitis within 1 year before informed consent or past medical history of chronic pancreatitis at time of informed consent.
15. Clinically significant heart disease at time of informed consent, including:

    1. History of documented congestive heart failure (New York Heart Association functional classification III-IV)
    2. Clinically significant uncontrolled cardiac arrhythmias
    3. Long QT syndrome, family history of idiopathic sudden death or congenital long QTsyndrome
    4. Corrected QT (QTcF) at screening: >470 ms for ≥18 years old / >450 ms for <18 years old
    5. Creatinine clearance < 70ml/min/1.73 m²
16. Patient currently, or in the 3 months before inclusion, enrolled in another interventional trial.
17. Person not affiliated to a national health insurance scheme
18. Patient, parents or legal authorized reprensentative incapable of expressing consent
19. Inability to attend all trial visits
20. For the optional consent only : contra indication to lumbar puncture:

    1. Known intracranial hypertension
    2. infection at puncture site
    3. known coagulation disorders
    4. Platelets < 50 × 109/L

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with response at end of treatment assessed by the Vineland II Adaptive Behavior Scale (VABS-II) | At 24 months of treatment compared to baseline
  Response defined by an improvement of at least 4 points in the Vineland II Adaptive Behavior Scale (VABS-II). The VABS-II consists of a form which will be filled during an interview with an adult who is familiar with the everyday activities of the patient (usually the parents). It is organized within a three-domain structure: communication, daily living skills, and socialization. In addition, VABS-II has a motor skills domain for the youngest children (younger than 6) and an optional maladaptive behavior index [Sparrow et al.,2016]. The domains (communication, daily living skills, and socialization) - standard scores have a mean of 100 and a standard deviation of 15. Adaptive levels can also be determined. A global standard score can also be computed (the Adaptive Behavior Composite standard score) and also has a mean of 100 and a standard deviation of 15.

SECONDARY OUTCOMES:
Proportion of patients randomized with a response (yes/no) in group A and group B | 6 months of treatment in double blind period
  Improvement of at least 4 points in the Vineland II Adaptive Behavior Scale (VABS-II) at 6 months of treatment in the group A compared to the group B
Changes from baseline in brain volume, vascularization, structural connectivity | baseline to end of treatment period
  Description of changes in brain volume, vascularization, structural connectivity, assessed by MRI
Frequency and severity of adverse events | Up to 34 months
  Type, frequency, seriousness, and severity of adverse events per CTCAE v5.0 criteria
Proportion of participants with response at end of treatment | At 6, 12 and 18 months of treatment, compared to baseline
  Improvement of at least 4 points in the Vineland II Adaptive Behavior Scale (VABS-II)
Change in quality of life assessed by Pediatric Quality of Life Inventory 4.0 or San Martin questionnaires | At 6, 12, 18, 24 months of treatment, compared to baseline.
  Pediatric Quality of Life Inventory 4.0 (PedSQL): The quality of life questionnaire PedSQL 4.0 consists of a modular approach to measuring health-related quality of life in healthy children and adolescents (ages range : 2-18 years). It is brief (23 items only). It takes less than 10 minutes to complete. This scale is designed to assess 4 dimensions: physical, emotional, social and school functioning. It is valid, reliable and sensitive to change.
  - The San Martin Scale is completed by parents or primary caregiver who knows well the person with ID, for at least three months. They have to rate each item on a 4-point scale (from 1= when the item is never true, to 4 = when it is always true). The questionnaire consists of 95 items, assessing eight dimensions of the quality of life
Evolution of scores at visual analogue scale | At 6, 12, 18, 24 months of treatment, compared to baseline.
Evolution of Clinical Global Impression of severity (CGI-S) | At 6, 12, 18, 24 months of treatment, compared to baseline.
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
Evolution of Global improvement scores (CGI-I) | At 6, 12, 18, 24 months of treatment, compared to baseline.
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention
Changes in neuropsychological scales adapted to age for attention, cognition, visuo-spatial disorders, fine motor skills, speech, reasoning and cognitive inhibition abilities | At 12 and 24 months of treatment compared to baseline
  Appropriate neuropsychological tests will be used according to the age of patients and their level of cognitive impairment. The tests were selected according to the conclusions of a working group from the DéfiScience Network (see link), which assessed all the neuropsychological tests available for each domain and adapted to ID patients, and the lack of sensitivity to placebo effect. In case of mild to moderate ID, appropriate Wechsler scale will be used. In case of severe ID, Revised-Brunet-Lézine scale will be used. Attention, visuo-spatial, language and fine motor skills will be assessed using subtests from Wechsler scales, NEPSY II and the Children Memory Scale or WMS IV for adults.
Changes in seizures frequency | At 6, 12, 18 and 24 months of treatment compared to baseline
  Evolution of number of epileptic seizures for affected patients and antiepileptic drugs use, assessed by a weekly diary
Changes in overgrowth or skin lesions | At 6, 12, 18 and 24 months of treatment compared to baseline
  Increase, no changes or reduction according to clinical measures and standardized photographs
Changes in Motor Function Measure (MFM) scores | At 6, 12, 18 and 24 months of treatment compared to baseline
  Motor Function Measure (MFM) is a comprehensive quantitative scale created to measure functional motor skills in a person with neuromuscular disease. It makes possible to classify patients in grade of severity in each of the 3 areas of motor function (D1: standing position and transfers, D2: axial and proximal motor skills, D3: distal motor skills).
Pharmacokinetic parameters of alpelisib (ng/mL) in cerebrospinal fluid (CSF) and blood | Between 6 and 24 months of treatment
  Level of alpelisib (ng/mL) in CSF and in blood, and correlation estimate (rho) between CSF and blood levels of alpelisib

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - CHRU Brest, Brest
  - HCL - Groupement Hospitalier Est Hôpital Femme-Mère-Enfant, Bron
  - Chu Estaing, Clermont-Ferrand
  - Chu Dijon Bourgogne, Dijon
  - CHU Dijon Bourgogne - CIC-P, Dijon
  - CHU de Lille, Lille
  - CHRU Nîmes, Nîmes
  - AP-HP Hôpital Necker-Enfants Malades - CIC, Paris
  - AP-HP Hôpital Necker-Enfants Malades, Paris
  - CHU Rennes, Rennes
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All requests for the study's data will be considered by the SESAM trial steering committee.

REFERENCES:
- [Background] Sparrow SSC, D.V.; Saulnier, C.A. Vineland-3: Vineland Adaptive Behavior Scales. 3rd ed. Pearson Assessments; Minneapolis, MN, USA. 2016.
- [Background] Curie A, Brun A, Cheylus A, Reboul A, Nazir T, Bussy G, Delange K, Paulignan Y, Mercier S, David A, Marignier S, Merle L, de Freminville B, Prieur F, Till M, Mortemousque I, Toutain A, Bieth E, Touraine R, Sanlaville D, Chelly J, Kong J, Ott D, Kassai B, Hadjikhani N, Gollub RL, des Portes V. A Novel Analog Reasoning Paradigm: New Insights in Intellectually Disabled Patients. PLoS One. 2016 Feb 26;11(2):e0149717. doi: 10.1371/journal.pone.0149717. eCollection 2016. PMID 26918704
- [Derived] Luu M, Vabres P, Espitalier A, Maurer A, Garde A, Racine C, Carpentier M, Rega A, Loffroy R, Hadouiri N, Boddaert N, Curie A, Guibaud L, Chebbi M, Charligny J, Kuentz P, Canaud G, Bahi-Buisson N, Fleck C, Cransac A, Bardou M, Faivre L; SESAM study group. A phase II double-blind multicentre, placebo-controlled trial to assess the efficacy and safety of alpelisib (BYL719) in paediatric and adult patients with Megalencephaly-CApillary malformation Polymicrogyria syndrome (MCAP): the SESAM study protocol. BMJ Open. 2024 Dec 20;14(12):e084614. doi: 10.1136/bmjopen-2024-084614. PMID 39806603
- See also: Related Info — http://www.defiscience.fr